CLINICAL TRIAL: NCT03083873
Title: A Phase 2, Multicenter Study to Evaluate the Efficacy and Safety of Autologous Tumor Infiltrating Lymphocytes (LN-145/LN-145-S1) for the Treatment of Patients With Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of LN-145/LN-145-S1 Autologous Tumor Infiltrating Lymphocytes in the Treatment of Squamous Cell Carcinoma of the Head & Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-145-03; 2016-003446-86 (EudraCT Number)
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: LN-145; Cell Therapy; Autologous Adoptive Cell Transfer; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; Tumor Infiltrating Lymphocytes; TIL; IL-2; LN-145-S1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Toll-Like Receptor 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Treatment with LN-145, Generation 1 (Gen 1), non-cryopreserved TIL
  Interventions: Biological: LN-145
- Cohort 2 (Experimental): Treatment with LN-145 Generation 2 (Gen 2), cryopreserved TIL
  Interventions: Biological: LN-145
- Cohort 3 (Experimental): Treatment with LN-145 Generation 3 (Gen 3), cryopreserved TIL
  Interventions: Biological: LN-145
- Cohort 4 (Experimental): Treatment with LN-145-S1 cryopreserved TIL
  Interventions: Biological: LN-145-S1
- Cohort 5 (Experimental): LN-145 cryopreserved/LN-145-S1 cryopreserved TIL re-treatment
  Interventions: Biological: LN-145; Biological: LN-145-S1

INTERVENTIONS:
Biological: LN-145 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After NMA lymphodepletion, patients are infused with their autologous TIL (LN-145) followed by IL-2 administration.
  Other Names: TIL, autologous tumor infiltrating lymphocytes
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 5
Biological: LN-145-S1 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After NMA lymphodepletion, patients are infused with autologous TIL (LN-145-S1) followed by IL-2 administration.
  Other Names: TIL, autologous tumor infiltrating lymphocytes
  Arms: Cohort 4; Cohort 5

SUMMARY:
Multicenter, multicohort, non-randomized, prospective, open label, interventional study evaluating adoptive cell therapy (ACT) with autologous tumor infiltrating lymphocytes (TIL) infusion (LN-145/LN-145-S1) followed by IL-2 after a non-myeloablative (NMA) lymphodepletion preparative regimen for the treatment of patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck

DETAILED DESCRIPTION:
LN-145/LN-145-S1 is an adoptive cell transfer therapy that utilizes an autologous TIL manufacturing process, as originally developed by the NCI, for the treatment of patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck. The cell transfer therapy used in this study involves patients receiving a NMA lymphodepletion preparative regimen, followed by infusion of autologous TIL followed by the administration of a regimen of IL-2.

ELIGIBILITY:
Inclusion Criteria

* Must be greater than 18 years of age at the time of consent.
* Must have recurrent and/or metastatic, squamous cell carcinoma of the head and neck (both HPV-positive and -negative)
* Must have at least 1 lesion that is resectable for TIL generation.
* Must have measurable disease as defined by RECIST v1.1 following the surgical resection.
* Must have received at least 1 and no more than 3 lines of prior systemic immunotherapy and/or chemotherapeutic treatments for HNSCC.
* Any prior therapy directed at the malignant tumor must be discontinued at least 28 days prior to lymphodepletion.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients must be seronegative for the human immunodeficiency virus.
* Patients seropositive for hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), or hepatitis C virus (anti-HCV) indicating acute or chronic infection may be enrolled if the viral load by polymerase chain reaction (PCR) is undetectable with/without active treatment
* Patients of childbearing potential and patients whose sexual partners are of childbearing potential must be willing to practice an approved method of highly effective birth control starting at the time of informed consent and for 1 year after the completion of the study treatment regimen.

Exclusion Criteria:

* Patients who have received an organ allograft or prior cell transfer therapy within the past 20 years.
* Patients who are on a systemic steroid therapy (greater than 10 mg of prednisone or equivalent). Patients receiving steroids as replacement therapy for adrenocortical insufficiency at < 10 mg of prednisone or other steroid equivalent daily may be eligible.
* Prior therapy-related toxicities Grade ≥ 1 according to Common Toxicity Criteria for Adverse Events (CTCAE) v4.03
* Patients with documented Grade ≥ 2 diarrhea or colitis as a result of previous immunotherapy within six months from screening.
* Patients who have a contraindication to or history of hypersensitivity reaction to cyclophosphamide, mesna, fludarabine, IL-2, antibiotics of the aminoglycoside group (ie, gentamicin or streptomycin; excluding those who are skin-test negative for gentamicin hypersensitivity), any component of the TIL infusion product formulation including dimethylsulfoxide (DMSO), human serum albumin (HSA), IL-2, and dextran-40.
* Patients with active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system.
* Patients with symptomatic and/or untreated brain metastases.
* Have any form of primary or acquired immunodeficiency syndrome, such as severe combined immunodeficiency disease or acquired immune deficiency syndrome (AIDS).
* Patients who have a left ventricular ejection fraction (LVEF) < 45% or who are New York Heart Association (NYHA) Class 2 or higher.
* Patients who have had another primary malignancy within the previous 3 years.
* Patients who are pregnant, parturient, or breastfeeding women.
* Patients who have received a live or attenuated vaccine within 28 days of the NMA-LD regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Medical Monitor, Study Director — Iovance Biotherapeutics
Locations (22):
- United States (22):
  - University of Alabama, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of Southern California, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Christiana Care Health System, Newark, Delaware
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Westwood, Kansas
  - University of Louisville, Louisville, Kentucky
  - Louisiana State University - Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - Providence Cancer Center Oncology and Hematology Care Clinic, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Washington, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Ferris RL MD,, Leidner RS, Chung CH, Jimeno A, Lee SM, Sukari A, Nieva JJ, Grilley-Olson JE, Redman R, Wong SJ, Villaflor VM, Misleh J, Finckenstein FG, Chou J, Gastman B, Fiaz R, Catlett M, Yi M, Cohen EEW. Efficacy and safety of one-time autologous tumor-infiltrating lymphocyte cell therapy in patients with recurrent and/or metastatic head and neck squamous cell carcinoma. J Immunother Cancer. 2025 Aug 24;13(8):e011633. doi: 10.1136/jitc-2025-011633. PMID 40854613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 20 centers that screened participants and 18 that enrolled participants in the United States, Jan 2017 through Aug 2022.
Pre-assignment Details: No participants were enrolled in Cohort 5 (TIL Retreatment Cohort) thus Cohort 5 (TIL Retreatment Cohort) has zero participants.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started (Enrolled / Tumor Harvested) | 10 | 22 | 19 | 13 | 0
Infused With TIL | 8 | 17 | 16 | 12 | 0
Completed Assessment Period (From TIL infusion on Day 0 and ends upon disease progression, the start of a new anticancer therapy, withdrawal of consent, or after 2 years (Month 24), whichever occurred first.) | 8 | 15 | 11 | 9 | 0
Completed (Completed 3 years after enrollment.) | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 22 | 19 | 13 | 0
Not completed — Death | 6 | 15 | 13 | 9 | 0
Not completed — Sponsor Terminated Study | 0 | 1 | 2 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0
Not completed — Did Not Receive TIL | 2 | 5 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set is defined as patients who have received LN-145/LN-145-S1 infusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 8 | 17 | 16 | 12 | 0 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 10 | 12 | 10 | 0 | 40
  >=65 years | 0 | 7 | 4 | 2 | 0 | 13
Age, Continuous [Median (Full Range); unit: years] | 57 [24 to 64] | 58 [37 to 71] | 56 [34 to 67] | 56.5 [50 to 75] |  | 57 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 |  | 7
  Male | 7 | 15 | 14 | 10 |  | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 |  | 3
  Not Hispanic or Latino | 7 | 17 | 14 | 10 |  | 48
  Unknown or Not Reported | 1 | 0 | 1 | 0 |  | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 |  | 0
  Asian | 0 | 0 | 0 | 2 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 1 | 1 | 1 |  | 3
  White | 8 | 16 | 15 | 9 |  | 48
  More than one race | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 17 | 16 | 12 |  | 53

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The percentage of patients who have a confirmed complete response or partial response as assessed by the investigator per RECIST v1.1. Objective response rate (ORR) will be defined as the percentage of the patients with a confirmed complete or partial response (CR or PR),by MRI or CT scan as per RECIST 1.1 criteria.
  Complete response (CR), Disappearance of all target and non-target lesions. All lymph nodes must be non-pathological in size(<10mm short axis). No new lesions.
  Partial response (PR), At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Persistence of one or more non-target lesion(s) and/or maintenance above the normal limits (Non-CR/Non-PD). No new lesions.
Time Frame: Up to 24 months
Population: The Full Analysis Set is defined as patients who have received LN-145/LN-145-S1 infusion that meets the manufacturing product specification.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 17 | 16 | 12
percentage of patients | 37.5 [8.5 to 75.5] | 5.9 [0.1 to 28.7] | 0 [0 to 20.6] | 16.7 [2.1 to 48.4]

2. Secondary Outcome: Duration of Response
Description: To evaluate efficacy parameters such as Duration of Response (DOR) using RECIST v1.1 as assessed by the Investigator. DOR is measured from the time point at which the initial measurement criteria per RECIST v1.1 are met for a CR or PR (if response is a confirmed response), whichever response is observed first, until PD.
Time Frame: Up to 24 months
Population: Participants who had confirmed responses from the Full Analysis Set. The Full Analysis Set is defined as patients who have received LN-145/LN-145-S1 infusion that meets the manufacturing product specification.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 3 | 1 | 0 | 2
Months | 3.1 [2.8 to 7.6] | NA [NA to NA] — Insufficient number of participants with events, therefore the Median and 95% Confidence Interval could not be calculated |  | NA [7.6 to NA] — Insufficient number of participants with events, therefore the Median and 95% Confidence Interval could not be calculated

3. Secondary Outcome: Disease Control Rate
Description: The percentage of patients who have a best overall response of complete response, partial response, or stable disease as assessed by the investigator per RECIST v1.1. The BOR of SD must be at least 4 weeks from LN-145/LN-145-S1 infusion.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 17 | 16 | 12
percentage of patients | 87.5 [47.3 to 99.7] | 70.6 [44.0 to 89.7] | 75.0 [47.6 to 92.7] | 75.0 [42.8 to 94.5]

4. Secondary Outcome: Progression-Free Survival
Description: The time (in months) from the date of the TIL infusion to progressive disease as assessed by the Investigator using RECIST v1.1 or death due to any cause, whichever occurs earlier. Progression was defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) as at least a 20% increase in the sum of diameters of the target lesions and an absolute increase of at least 5 mm, and/or unequivocal progression of existing non-target lesions, and/or the appearance of 1 or more new lesions.
Time Frame: Up to 24 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 8 | 17 | 16 | 12
Months | 2.8 [0.9 to 3.9] | 1.9 [1.6 to 2.8] | 2.8 [1.8 to 3.1] | 1.9 [0.6 to 9.0]

ADVERSE EVENTS:
Time Frame: 5 years, 5 months
Description: Treatment-emergent adverse events (TEAEs), clinical laboratory data assessments, serious adverse events (SAEs), and adverse events (AEs) were collected and evaluated for the duration of the study until resolution or permanent sequelae. The Safety Analysis Set is defined as patients who have received TIL infusion.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 6/8 | 15/17 | 13/16 | 9/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/8 | 9/17 | 11/16 | 8/12 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 17/17 | 16/16 | 12/12 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=17) | Cohort 3 (N=16) | Cohort 4 (N=12) | Cohort 5 (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 2 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia [1] (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Thrombocytopenia [2] (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Capillary leak syndrome (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 3 | 2 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=8) | Cohort 2 (N=17) | Cohort 3 (N=16) | Cohort 4 (N=12) | Cohort 5 (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 | 7 | 9 | 8 | 0
Basophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 5 | 5 | 0
Leukopenia [1] (Blood and lymphatic system disorders) | 3 | 6 | 5 | 5 | 0
Lymphopenia [2] (Blood and lymphatic system disorders) | 4 | 5 | 2 | 2 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia [3] (Blood and lymphatic system disorders) | 3 | 5 | 5 | 6 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia [4] (Blood and lymphatic system disorders) | 4 | 12 | 12 | 10 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 2 | 2 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 3 | 1 | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 7 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 4 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 1 | 0
Chills (General disorders) | 6 | 12 | 7 | 7 | 0
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 3 | 2 | 0
Hypothermia (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Mass (General disorders) | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 1 | 4 | 0
Pain (General disorders) | 0 | 2 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 5 | 10 | 7 | 4 | 0
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 3 | 2 | 0
Scrotal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 3 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood culture positive (Investigations) | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 1 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 1 | 2 | 0
Weight increased (Investigations) | 1 | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5 | 4 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 5 | 8 | 3 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 4 | 5 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 7 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 5 | 3 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 6 | 9 | 3 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 2 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 3 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2 | 3 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 5 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 4 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Cyanosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Distributive shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 2 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 3 | 3 | 0
Hypotension (Vascular disorders) | 5 | 6 | 7 | 7 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor's agreements with sites ensure the site/investigator may publish study results following the earlier of a multicenter publication or 18 months after end of the multicenter trial consistent with academic standards for non-commercial purposes. Sponsor may review the publication for 30-60 days to remove confidential information and up to 60-90 more days to protect its intellectual property. Sponsor may not prohibit disclosure of site's results.

DOCUMENTS (5):
  • Study Protocol: Version 1 (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT03083873/Prot_000.pdf
  • Study Protocol: Version 2 (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT03083873/Prot_001.pdf
  • Study Protocol: Version 3 (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT03083873/Prot_002.pdf
  • Study Protocol: Version 4 (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT03083873/Prot_003.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03083873/SAP_004.pdf